CLINICAL TRIAL: NCT01447966
Title: Family Based Cognitive-Behavioral Treatment for Preschoolers With Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Adam Lewin, Assistant Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YC-OCD
Record Dates: First submitted 2011-09-29; First posted 2011-10-06 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: OCD; Obsessive Compulsive Disorder; Child; Pediatric; CBT; Therapy; ERP; Exposure Response Prevention; Preschool; Cognitive Behavioral
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as Usual (No Intervention): Participants randomized to the TAU arm will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions). Treatment changes (e.g., medication increase, starting psychotherapy in the community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice.
- Immediate CBT (Experimental): Therapists will work with families for 12 twice weekly sessions, each lasting up to 60 minutes implementing a developmentally appropriate modulated cognitive behavioral therapy approach. A manualized CBT protocol will be followed.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Family based cognitive behavioral therapy with exposure and response prevention. Twice weekly for 45-60 minute visits.
  Other Names: ERP - Exposure response prevention
  Arms: Immediate CBT

SUMMARY:
The purpose of this research study is to further investigate how well cognitive-behavioral psychotherapy works to reduce obsessive-compulsive symptoms in young children with obsessive-compulsive disorder (OCD). Cognitive-behavioral therapy has been shown to work well in youth with OCD and other anxiety disorders; however, there are only a few studies to date in preschool and young children with OCD. All children will have the option to receive 12 twice-weekly cognitive-behavioral psychotherapy sessions that are up to 60-minutes each. Randomly determined, half of all children will receive these sessions immediately following the pre-assessment and the remaining half will receive them after six weeks. The investigators expect that youth receiving the study-based therapy will show more improvement in OCD symptoms in six weeks in contrast to youth waiting to receive the therapy.

DETAILED DESCRIPTION:
Cognitive Behavioral Therapy for OCD includes several core therapeutic elements including establishment of treatment goals, assigned homework, operant conditioning paradigms (the putative mechanism for exposure-based therapies), provision of psychoeducation (e.g., the link between thoughts, feelings, and behaviors), cognitive (e.g., cognitive restructuring) and behavioral (e.g., exposure) coping skill implementation, and target behavior progress assessments. Nevertheless, research is lacking in preschoolers with OCD and these children likely require adaptations to the traditional CBT regimen. Preschoolers often have a high level of family accommodation, whereby the family members become part of the rituals and compulsions in attempt to ease the young child's anxiety. CBT with preschoolers will need to emphasize delivering intervention within the context of the family. The flexibility of this modular approach for treatment (modular therapies allow for variations in the order and intensiveness of the aforementioned treatment elements, providing an individually tailored treatment instead of a one-size-fits-all approach) may be optimally suited for preschoolers with OCD given their wide variability in developmental level and symptom presentation. This is consistent with the NIH Roadmap Initiative which calls for personalized interventions matched to individual patient characteristics. Our OCD research team in the Rothman Center is highly experienced in clinical research for pediatric and adult OCD. The proposed investigation is a single-site controlled trial of CBT in preschool aged youth with OCD aged 3-8 years. We will randomly assign patients to immediate treatment or 6-week Treatment as Usual (TAU) control. A manualized CBT protocol will be followed. Assessments will occur at Screening, Baseline, Post-treatment and 1 and 3-month follow-ups. Ratings of patient OCD symptom severity will be conducted at each time point by trained raters blinded to treatment condition. Diagnosis will be established by an experienced clinician and verified by a validated rating scale conducted with the child's parent(s); cases will be reviewed by study investigators. Assessments will be audio-recorded and verified for integrity. Randomization will be determined immediately following the baseline assessment; patients will be assigned TAU or immediate treatment in a 1:1 ratio. All eligible patients will receive 12 therapy sessions over 6 weeks using the evidence-based treatment protocol that incorporates E/RP and parent involvement; sessions are twice weekly for 60 minutes. Dr. Lewin and other trained OCD therapists under his supervision will conduct therapy sessions. All sessions are audiorecorded for integrity.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV-TR for a primary diagnosis of OCD
* Minimum score of 8 on the CYBOCS compulsion scale
* Peabody Picture Vocabulary IV score of 80
* Able to attend biweekly appointments with a parent/guardian
* English Speaking

Exclusion Criteria:

* Current clinically significant suicidality
* engaged in suicidal behaviors within 6 months
* Peabody Picture Vocabulary IV score of 80
* Any change in established psychotropic medication (e.g., antidepressants, anxiolytics) within 4 weeks before study enrollment, any change in antipsychotics within 3 weeks prior to the screening assessment, any change in Prozac or Straterra within 6 weeks of study enrollment, and any change in alpha-2 agonists or stimulants within 1 week of study enrollment.
* Lifetime DSM-IV bipolar, schizophrenia or schizoaffective disorders; or Substance abuse in past 6 months.
* Absence of language
* Formal diagnosis of mental retardation or an autism spectrum disorder
* Unwillingness of parents to make the commitment to accompany their child for multiple study visits, unwillingness to take part in randomization, inability to attend sessions twice weekly as therapist availability allows, inability to attend assessment visits.
* Presence of a significant and/or unstable medical illness which might lead to hospitalization during the study.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2011-05; Primary Completion 2013-06 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Clinician Global Impression - Improvement Scale (Measure of patient improvement at relevent timepoints) | Baseline/Post-treatment or Post-waitlist/1 and 3 Month Follow-up
  The CGI is a 7-point rating of treatment response anchored by 1 ("very much improved), 4 ("no change") and 7 ("very much worse"). Youth being rated by the IE as 1 ("very much improved") and 2 ("much improved") will be considered treatment responders. This measure assesses change or improvement across time and consequently is appropriate for use at multiple assessments - reflects patient improvement relative to baseline functioning. Represents change in functioning and assesses change in baseline. Appropriate for use at multiple time-points.

SECONDARY OUTCOMES:
CYBOCS - Childrens Yale Brown Obsessive Compulsive Scale | Baseline, post-treatment/post waitlist, 1 and 3 month followup
  The CY-BOCS is a 10-item semi-structured measure of obsession and compulsion severity over the previous week. Measure will be administered to the parent.
  Change score (calculated as a percent change from baseline) will be used as the outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Adam B Lewin, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- University of South Florida - Rothman Center for Neuropsychiatry, St. Petersburg, Florida, United States

REFERENCES:
- [Derived] Lewin AB, Park JM, Jones AM, Crawford EA, De Nadai AS, Menzel J, Arnold EB, Murphy TK, Storch EA. Family-based exposure and response prevention therapy for preschool-aged children with obsessive-compulsive disorder: a pilot randomized controlled trial. Behav Res Ther. 2014 May;56:30-8. doi: 10.1016/j.brat.2014.02.001. Epub 2014 Mar 2. PMID 24657310